CLINICAL TRIAL: NCT00494364
Title: Gas Supply, Demand and Middle Ear Gas Balance: Sp Aim 3a Pt ii
Brief Title: Gas Supply, Demand and Middle Ear Gas Balance: Specific Aim 3a Part ii
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, J. Douglas Swarts, Associate Professor, University of Pittsburgh
Other Study IDs: PRO07040059; NIH P50DC007667
Record Dates: First submitted 2007-06-28; First posted 2007-06-29 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Healthy
Keywords: ear disease; otitis; Eustachian tube; mastoid air cells; Normal healthy volunteers
MeSH Terms: conditions — Ear Diseases; Otitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The middle ear is an airspace located behind the eardrum that consists of two connecting compartments. The compartment directly behind the eardrum is called the tympanum and contains the three small bones of the middle ear, the hammer, anvil and stapes, that function to transfer eardrum movements to the inner ear so that you can hear. Behind the tympanum is the mastoid cavity which is a larger airspace subdivided into small air cells of unknown function. For normal hearing, it is important that the air pressure in the middle ear is similar to that of the environment so that the eardrum can move freely in response to sounds. The air pressure of the environment is not constant and is affected by changes in weather conditions (high and low pressure systems that move through the area) and by changes in elevation above sea level (the fullness in your ears that can be noticed when you ride in an elevator or in an airplane). The air pressure in the middle ear also changes because middle ear gas is constantly leaking from that airspace to the blood that flows through the walls of the middle ear. These effects (changing environmental air pressures and changing middle ear air pressure) are independent and cause the middle ear and environmental pressures to be different from each other. Periodically and during swallowing or yawning, any existing difference between middle ear and environmental air pressure is reset to zero by the opening of a biological tube (the Eustachian tube) that connects the middle ear to the back of the nose. This allows gas flow between the middle ear and the environment which increases or decreases middle ear pressure to the level in the environment at that time. Most people cannot open their Eustachian tubes at will and the number of automatic openings varies from infrequent to often in a population. Whether or not a person's usual frequency of Eustachian openings is good enough to keep the middle ear pressure the same as environmental levels depends on how fast gas is lost from the middle ear by gas leakage (diffusion) to blood. For example, in ears with very slow rates of gas loss, the Eustachian tube does not need to open very frequently to keep the middle ear at environmental pressure. Some researchers believe that the mastoid compartment functions to control the rate of gas loss to blood, with larger mastoid volumes associated with lesser rates of middle ear gas loss. In this experiment, the investigators plan to test this by measuring mastoid and tympanum volumes using Computer tomography (CT) and the rate of blood to middle ear gas transfer using a technique that involves breathing air that contains laughing gas (Nitrous Oxide=N2O) and measuring middle ear pressure change using tympanometry (a technique that involves putting an ear plug into the ear canal and measuring the pressure). From past studies in patients undergoing short surgical or dental procedures, the investigators know that breathing gas mixtures that contain N2O will increase the blood levels of that gas, cause gas to go from blood to the middle ear and increase middle ear pressure. The investigators predict that the rate of change in middle ear pressure while breathing a gas mixture containing 25% N2O and the normal oxygen level (20%) of air will be less for those ears with larger mastoid volumes. If the investigators prediction is correct, they will be able to explain why ears with larger mastoid volumes are better able to keep their pressure like that of the environment even if the Eustachian tube does not open often.

DETAILED DESCRIPTION:
The middle ear (ME) pressure balance is an important contributor to the maintenance of ME health. ME pressure is a measure of the number of contained gas moles and processes that add or remove gas moles from the relatively fixed volume ME cavity change its pressure. Three routes for ME gas exchange have been identified; 1) passive, gradient-dependent species exchange with the local blood via diffusion across the ME mucosa; 2) passive, gradient-dependent species exchange with the ambient environment via diffusion across the tympanic membrane, and 3) bolus exchange of mixed gases between the nasopharynx and ME during transient openings of the Eustachian tube. Total ME pressure and the trajectory of ME pressure under specified conditions depend on the relative rates of species gas exchanges across these pathways. The ME airspace can be subdivided into two compartments, the anterior tympanum and the posterior mastoid air cell system (MACS). Theory suggests that the transmucosal gas exchange rate for the ME (transMEM) may be different for the tympanum and the MACS and this possibility has important implications with respect to the role of the MACS in ME pressure regulation and protection from ME disease. This study measures the rate of inert gas exchange across the mucosa of the two ME compartments in adults. These data will be fitted to a model of gas exchange parameterized based on the relative surface areas and volumes of the two compartments, and the hypothesis that volume gas exchange across the MACS mucosa is less than that for the tympanum will be tested. The results will be used to reject or confirm one mechanism by which large MACS volume protects from otitis media under certain conditions.

ELIGIBILITY:
Inclusion Criteria:

* Both ears-drums intact and effusion-free

Exclusion Criteria:

* Chronic illness including asthma, lung, or heart disease
* Pregnant or plans on becoming pregnant during study period
* Prescription meds other than birth control
* Previous problems with inhaling nitrous oxide (e.g., during dental procedure)
* Claustrophobia in confined spaces
* Unable to remain relaxed and quiet for up to 2 hours

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adult volunteers
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2007-06; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William J Doyle, PhD, Principal Investigator — University of Pittsburgh; J. Douglas Swarts, PhD, Study Director — University of Pittsburgh
Locations (1):
- ENT Research Center, Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States